CLINICAL TRIAL: NCT07227506
Title: Diagnostic Utility of Mucosal Impedance Device in Patients With GERD and Chronic Esophageal Disorders:
Brief Title: Utility of Mucosal Impedance Device in Chronic Esophageal Disorders:
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Gokulakrishnan Balasubramanian, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00055595
Record Dates: First submitted 2025-11-11; First posted 2025-11-12 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Gerd; Eosinophilic Esophagitis
Keywords: gerd; eosinophilic esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- True GERD: Positive endoscopy findings or esophageal pH results based on Lyon 2.0
  Interventions: Device: MuVI Esophageal mucosal impedance testing
- Functional Heartburn: Negative endoscopy and negative esophageal pH testing results
  Interventions: Device: MuVI Esophageal mucosal impedance testing

INTERVENTIONS:
Device: MuVI Esophageal mucosal impedance testing — Esophageal mucosal impedance values are checked in both groups

SUMMARY:
Background & Significance Chronic benign esophageal disorders such as Gastroesophageal reflux disease (GERD) and eosinophilic esophagitis are common gastrointestinal disorders affecting nearly 20% and 0.1% of the population, respectively. Although these conditions are frequent, the diagnosis of GERD or EoE requires complex decision making involving endoscopic examination, histopathological examination, and esophageal pH testing. This translates into significant economic burden; For example, burden due to GERD is about $24 billion annually. Additionally, there may be a delay in the diagnosis of GERD or EoE as Investigators might have to do multiple procedures such as upper endoscopy, esophageal pH testing, etc for the same participant for confirmation of the diagnosis. In addition, there could be overlay between GERD and EoE in the diagnosis which make cause delay in the diagnosis and decision making.

Aim:

Here, Investigators will plan to identify the diagnostic utility and cost-effectiveness of this novel Mivu device(FDA approved) in the diagnosis of gastroesophageal reflux disease or chronic esophageal inflammatory disorders in participants with reflux symptoms or chronic esophageal symptoms.

DETAILED DESCRIPTION:
Diagnostic Utility of Mucosal Impedance Device in participants with GERD and chronic esophageal disorders:

Background & Significance Chronic benign esophageal disorders such as Gastroesophageal reflux disease (GERD) and eosinophilic esophagitis are common gastrointestinal disorders affecting nearly 20% and 0.1% of the population, respectively. Although these conditions are frequent, the diagnosis of GERD or EoE requires complex decision making involving endoscopic examination, histopathological examination, and esophageal pH testing. This translates into significant economic burden; For example, burden due to GERD is about $24 billion annually. Additionally, there may be a delay in the diagnosis of GERD or EoE as Investigators might have to do multiple procedures such as upper endoscopy, esophageal pH testing, etc for the same participant for confirmation of the diagnosis. In addition, there could be overlay between GERD and EoE in the diagnosis which make cause delay in the diagnosis and decision making.

In summary, current diagnostic testing for GERD lead to several challenges:

* Delayed diagnosis, particularly in cases where participants undergo normal endoscopy but still experience symptoms.
* Increased healthcare costs, with GERD alone accounting for an estimated $24 billion annually in the United States.
* Diagnostic overlap between GERD and EoE, which complicates clinical decision-making and contributes to further delays or misdiagnoses.

Since majority of the participants who undergo upper endoscopy for GERD, have normal endoscopic visualization of esophagus, esophageal pH impedance or wireless pH testing are essential to make the diagnosis of GERD. Hence, Esophageal Mucosal impedance (Mivu) is a measurement tool that can evaluate if the structure of the esophageal mucosal tissue as a one-stop solution testing. MI is performed using an FDA approved endoscopic tool called "Mucosal Integrity Conductivity Test System" (Diversatek). The Mivu system software uses the collected data to determine if there is evidence of GERD.

Prior studies have demonstrated a positive correlation between low mucosal impedance and conditions such as GERD and EoE. As such, Mivu offers the potential to:

* Serve as a single-procedure diagnostic approach.
* Reduce diagnostic delay and resource utilization.
* Improve accuracy in differentiating between GERD, EoE, and functional heartburn.

Aim:

Here, Investigators will plan to identify the diagnostic utility and cost-effectiveness of this novel Mivu device(FDA approved) in the diagnosis of gastroesophageal reflux disease or chronic esophageal inflammatory disorders in participants with reflux symptoms or chronic esophageal symptoms.

Methods:

Study:

This is a prospective study aimed at evaluating chronic benign esophageal disorders such as gastroesophageal reflux disease and eosinophilic esophagitis. All the participants with reflux symptoms or dysphagia/esophageal symptoms who undergo upper endoscopy will be enrolled into the study.

Step by Step Procedure:

1. During routine esophagogastroduodenoscopy (EGD) visit, consented study participants will be given GERD questionnaire.
2. During endoscopic evaluation of the esophagus as a part of standard of care, Investigators will make sure there is no esophageal stricture or malignancy.
3. Subsequently, original single channel Mivu catheter (FDA approved) advanced to the distal esophagus.
4. Measurements of mucosal impedance will be taken at proximal, mid and distal esophageal locations for 5 seconds each.
5. Once the mucosal impedance data have been recorded, the assembly will be deflated and removed by the investigator.
6. The study procedure will add approximately 1-5 minutes of procedure time for each research participant.
7. Participants will undergo further diagnostic testing as per standard of care.
8. Those participants who are diagnosed with Grade C or D esophagitis at the initial visit will return for a follow-up visit after treatment with proton pump inhibitor (PPI) therapy to determine whether or not esophagitis has healed as part of their standard of care.

Clinical Parameters that will be collected:

Clinical:

1. Demographics (age, sex, race, and body mass index).
2. GERD questionnaire.
3. Dysphagia symptom severity using Mayo Dysphagia Scale and hypervigilance questionnaire.

Endoscopic:

1. Presence and size of a hiatal hernia.
2. Presence and severity of esophagitis (graded by the Los Angeles Classification: A, B, C, or D).
3. Novel Mucosal impedance data: proximal and distal esophageal sensor.
4. Endoflip data if done as part of standard of care- esophageal distensibility index.
5. Standard esophageal pH and impedance testing if done as part of standard of care: Proximal and distal acid exposure times over the study period, nocturnal basal impedance.
6. Pathology Data if done as part of standard of care: Eosinophil count (proximal and distal esophageal counts).
7. Esophageal manometry if done as part of standard of care: esophageal contractility integral, relaxation of lower esophageal sphincters.

Clinical Outcomes:

1. Diagnostic utility of mucosal impedance in the diagnosis of GERD; correlation of esophageal pH parameters with mucosal impedance data.
2. Cost-effectiveness of Mivu compared to the standard diagnostic testing tools such as esophageal pH or Bravo testing.
3. Correlation of esophageal inflammation in benign esophageal inflammatory disorders such as eosinophilic esophagitis and mucosal impedance values from Mivu.

Analysis:

This study will compare questionnaire scores and mucosal impedance scores in participants with GERD. All the categorical and numerical variables will be compared by Fischer's exact and Mann-Whitney test, respectively. Diagnostic utility (sensitivity and specificity of the new Mivu device will be calculated against the gold standard- endoscopy and esophageal pH testing. Sample size calculation after initial data collection of 50 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic esophageal symptoms such as atypical or typical reflux symptoms and dysphagia, is here for upper endoscopy testing.

Exclusion Criteria:

1. Presence of esophageal stricture
2. Unstable patients who cannot undergo this testing.
3. Patients on anticoagulation on the day of procedure.
4. Presence of esophageal cancer.
5. Pregnancy.
6. Minor patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the patients with reflux symptoms or dysphagia/esophageal symptoms who undergo upper endoscopy will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of MuVI | 1 year
  Sensitivity and Specificity of MuVI
Diagnostic utility of mucosal impedance in the diagnosis of GERD | 1 year
  Correlation of esophageal pH parameters with mucosal impedance data.

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not shared as per IRB policy due to potential HIPAA violation

REFERENCES:
- [Result] Choksi Y, Lal P, Slaughter JC, Sharda R, Parnell J, Higginbotham T, Vaezi MF. Esophageal Mucosal Impedance Patterns Discriminate Patients With Eosinophilic Esophagitis From Patients With GERD. Clin Gastroenterol Hepatol. 2018 May;16(5):664-671.e1. doi: 10.1016/j.cgh.2017.12.020. Epub 2017 Dec 14. PMID 29248733
- [Result] Patel DA, Higginbotham T, Slaughter JC, Aslam M, Yuksel E, Katzka D, Gyawali CP, Mashi M, Pandolfino J, Vaezi MF. Development and Validation of a Mucosal Impedance Contour Analysis System to Distinguish Esophageal Disorders. Gastroenterology. 2019 May;156(6):1617-1626.e1. doi: 10.1053/j.gastro.2019.01.253. Epub 2019 Jan 31. PMID 30711626
- [Result] Maresova P, Rezny L, Hruska J, Klimova B, Swanstrom LL, Kuca K. Diagnosis and treatment of patients with gastroesophageal reflux disease - a systematic review of cost-effectiveness and economic burden. BMC Health Serv Res. 2024 Nov 6;24(1):1351. doi: 10.1186/s12913-024-11781-8. PMID 39501242